CLINICAL TRIAL: NCT02490501
Title: An Open, Randomized, Rehabilitation-controlled Study to Assess Safety, Tolerability, and Efficacy of Heparin Activated Recombinant Fibroblast Growth Factor 1 on a Biodegradable Device in Subjects With Traumatic Spinal Cord Injury
Brief Title: Safety and Efficacy of SC0806 (Fibroblast Growth Factor 1 and a Device) in Traumatic Spinal Cord Injury Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioArctic AB (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC0806-A101
Record Dates: First submitted 2015-06-30; First posted 2015-07-03 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SC0806 (Active Comparator): Intervention with SC0806 (implantation of device with FGF1 and peripheral nerves) in addition to rehabilitation
  Interventions: Procedure: SC0806 and rehabilitation
- Controls (Other): Rehabilitation only
  Interventions: Other: Rehabilitation only

INTERVENTIONS:
Procedure: SC0806 and rehabilitation
  Arms: SC0806
Other: Rehabilitation only
  Arms: Controls

SUMMARY:
This is an open, randomized, rehabilitation-controlled study in subjects with complete Traumatic Spinal Cord Injury, where the active treatment consists of a surgical implantation of SC0806 (a biodegradable device with heparin-activated FGF1 and nerve implants).

DETAILED DESCRIPTION:
The study is a single dose study in up to 3 sequences in subjects with complete Traumatic Spinal Cord Injury. In each sequence, 6 subjects will be randomized to a surgical procedure where SC0806 will be implanted into the spinal cord and receive specific walking training, and 3 subjects will be randomized to specific walking training only. Interim analyses of safety parameters will be performed. If a positive effect and no major safety concerns have been demonstrated after completion of all sequences, the control subjects will be given the opportunity to receive treatment with SC0806 after completion of their rehabilitation periods.

ELIGIBILITY:
Inclusion Criteria:

1. Traumatic Spinal Cord Injury.
2. Male or female subjects aged between 18 and 65 years.
3. BMI ≤35, body weight ≤125 kg and height ≤ 195 cm at Screening.
4. Complete SCI (ASIA Impairment Scale level A, no voluntary bladder function, negative motor and sensory evoked potentials).
5. A single spinal cord lesion injury at the neurologic level between T2-T11.
6. A Baseline MRI that indicates a pathology consistent with a traumatic SCI
7. Minimum of 4 months and maximum 10 years post injury with no evidence of neurological improvement prior to implantation surgery unless there is a complete anatomical cut-off of the spinal cord.
8. Females must not be lactating or pregnant at Screening and Baseline (as documented by pregnancy tests).
9. All females that are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
10. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days before study entry and must agree to use a highly effective method of contraception (e.g., total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period. If currently abstinent, the subject must agree to use an effective method as described above if she becomes sexually active during the study period. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and must continue to use the same contraceptive during the study.
11. Written informed consent obtained prior to any study specific procedures.
12. Eligible for surgery and specific walking training as judged by the investigator.

Exclusion Criteria:

1. Other life-threatening injury.
2. Serious co-existing medical condition or mental disorder.
3. Results from neurophysiological examination preoperatively are inconsistent with a spinal cord injury of one thoracic segment or less.
4. Current or prior (within the past 8 weeks or within 5 half-lives of use of such a medication prior to screening) participation in any other investigational medication or device trial.
5. Known hypersensitivity to FGF1 or heparin.
6. Subjects unable to tolerate or undergo MRI scanning, including subjects with claustrophobia unless sedation can be used, cardiac pacemaker/defibrillator, ferromagnetic metal implants e.g., in skull, cardiac devices, other than those approved as safe for use in MR scanners.
7. Ongoing drug or alcohol abuse or dependence.
8. Positive serology for Hepatitis B or C, or Human Immunodeficiency Virus (HIV) at Screening.
9. Positive test for Methicillin-resistent Staphylococcus Aureus (MRSA) at screening.
10. Any disease, concomitant injury, condition or treatment that interferes with the specific walking training, the performance or interpretation of the neurological examination.
11. Has a condition or has received medical treatment that, in the judgment of the investigator, precludes successful participation in the study.
12. Previous radiation treatment (e.g. cancer treatment) in the region of the spinal cord injury.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06; Primary Completion 2020-10 (Actual); Study Completion 2025-05 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with an Adverse Event | 0 - 18 months
Proportion of subjects with an improvement, in the Motor Evoked Potential (MEP) scores | 0 - 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Hans Basun, MD, Study Director — BioArctic AB
Locations (1):
- Karolinska University Hospital and RSS, Stockholm, Sweden

REFERENCES:
- See also: Homepage of sponsor — http://www.bioarctic.se